CLINICAL TRIAL: NCT01134978
Title: Neural Mechanisms of the Contextual Interference Effect: A fNIRs and EEG Study
Acronym: GRID12007
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Drexel University (Other)
Collaborators: Pennsylvania Department of Health (Other Government)
Responsible Party: Patricia A. Shewokis, PhD, Drexel University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 16758
Record Dates: First submitted 2010-05-27; First posted 2010-06-02 (Estimated); Last update posted 2011-11-07 (Estimated); Status verified 2011-05

CONDITIONS: Healthy Individuals; Learning
Keywords: repeated measures design; random assignment to groups

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (1):
- Practice Schedules (Experimental): Subjects are randomly assigned to either a blocked or random practice schedule when learning three 3-D computer mazes. A blocked practice schedule is created when the tasks to be learned are presented in a predictable order, while a random practice schedule has tasks presented in a nonsequential, unpredictable order. Neural activity and behavioral measures will differ for the two practice schedules. For memory and transfer, it is predicted that random practice will be better than blocked practice.
  Interventions: Behavioral: Practice Order

INTERVENTIONS:
Behavioral: Practice Order — Blocked order - predictable
  Random order - unpredictable
  Other Names: High contextual interference - random practice schedule; Low contextual interference - blocked practice schedule

SUMMARY:
The overall goal of this study is to gain insight into the neural mechanisms of learning multiple tasks. By examination of cognitive and behavioral output during the performance and learning of several computer maze tasks, and through a detailed examination of the neural activity obtained from functional near-infrared (fNIR) and electroencephalography (EEG), it may be possible to gain insight into the impact of the amount of practice and the organization of practice has on learning fine motor skills. This insight may provide direction as to how to better develop instructional and rehabilitation protocols in addition to clinical interventions to facilitate recovery of function, relearning and transfer of cognitive and fine motor skills based upon neural responses to physical practice.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 55 years of age
* vision correctable to 20/20
* right-handed
* English is first language or learned English before age of 5 years

Exclusion Criteria:

* 17 years or younger and 56 years or older
* pregnant
* have latex or tape adhesives allergies
* self-exclude if:
* had a history of seizures, head injury or neurological dysfunction
* history or diagnosis of depression, schizophrenia or social phobia
* previous admission to alcohol/drug treatment program or diagnosis of alcohol/drug abuse
* take medications know to affect neurological function.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2007-11; Primary Completion 2010-12 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
metabolic measures of neural activity in the dorsolateral prefrontal cortex | outcomes measured 72 - 96 hours post-training
  Functional near infrared spectroscopy (fNIR) uses specific wavelets of light, that are introduced at the scalp to measure changes in the relative ratios of deoxygenated hemoglobin and oxygenated hemoglobin in the capillary beds during brain activity.

SECONDARY OUTCOMES:
Behavioral measures | measured 72-96 hours post training
  maze behavioral responses of time to traverse the maze (sec), distance traveled (pixels)and average maze velocity (pixels/sec) are calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Patricia A Shewokis, PhD, Principal Investigator — Drexel University
Locations (1):
- Cognitive Motor Movement Neuroscience Lab (CoMMoNS) - rm 3612 NCB, Drexel University, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Result] Ayaz H, Shewokis PA, Curtin A, Izzetoglu M, Izzetoglu K, Onaral B. Using MazeSuite and functional near infrared spectroscopy to study learning in spatial navigation. J Vis Exp. 2011 Oct 8;(56):3443. doi: 10.3791/3443. PMID 22005455
- [Result] Shewokis PA, Ayaz H, Izzetoglu M, Bunce S, Gentili RJ, Sela I, Izzetoglu K, Onaral B. Brain in the Loop: Assessing Learning using fNIR in cognitive and motor tasks. D.D. Schmorrow and C.M. Fidopiastis (Eds.).Lecture Notes in Artificial Intelligence, 6780: 240-249. 2011. Springer-Verlag Berlin Heidelberg 2011.
- [Result] Shewokis PA, Ayaz H, Izzetoglu K, Izzetoglu M, Bunce SC, Schultheis MT, Pourrezaei K. Dorsolateral prefrontal cortex activity during the learning of computer tasks in a contextual interference paradigm using fNIRs: a case series. Journal of Sport & Exercise Psychology 30: S130. 2008.
- [Result] Shewokis PA, Ayaz H, Izzetoglu M, Getchell N, Izzetoglu K. the acquisition and learning of computer tasks in a contextual interference paradigm: Using functional near infrared spectroscopy to examine prefrontal cortex activity. Journal of Sport & Exercise Psychology. 32: S127-S128. 2010.